CLINICAL TRIAL: NCT00585000
Title: A Phase 1, Open Label, Single Arm Study To Establish The Safety Of Administering CP 675,206 As A One Hour Infusion In Patients With Surgically Incurable Stage III Or Stage IV Melanoma
Brief Title: A Study To Assess The Safety Of Administering CP-675,206 As A One Hour Infusion In Patients With Surgically Incurable Advanced Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3671022
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: CP-675,206

INTERVENTIONS:
Drug: CP-675,206 — 15 mg/kg. IV (in the vein) over 1 hour on Day 1 of each 90 day cycle. Number of cycles: maximum of 4 cycles unless progression of disease or unacceptable toxicity.

SUMMARY:
This will show if CP-675,206 can be administered safely as an intravenous infusion lasting one hour. CP 675,206 already has been administered to 835 subjects over 1.0 - 7.5 hours.

DETAILED DESCRIPTION:
This study was prematurely discontinued on April 28, 2008 because a concomitant Phase 3 study met pre-specified futility criteria. The decision to close enrollment early was not based on any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed melanoma that is surgically incurable Note: Prior therapies for melanoma, including cancer vaccines, are permitted but are not required. There is no limit to the number of prior regimens for melanoma a patient may have received.
* Evidence of at least one lesion
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* CT scan of the brain with contrast or MRI of the brain within 6 weeks prior to enrollment showing no evidence of active brain metastases. PET scans and PET/CT scans are also acceptable.

Exclusion Criteria:

* Previous treatment with other anti CTLA4 agents (eg, ipilimumab, MDX 010).
* Previously randomized to Pfizer study A3671009: A Phase 3, Open Label, Randomized Comparative Study of CP 675,206 and Either Dacarbazine or Temozolomide in Patients with Advanced Melanoma.
* History of chronic autoimmune disease (eg, Addison's disease, multiple sclerosis, Graves disease, Hashimoto's thyroiditis, psoriasis, rheumatoid arthritis, systemic lupus erythematosus, hypophysitis, etc.).
* History of inflammatory bowel disease (eg, Crohn's disease or ulcerative colitis), celiac disease, or other chronic gastrointestinal conditions associated with diarrhea, or current acute colitis of any origin, and any history of diverticulitis (even a single episode) or evidence of diverticulitis at baseline, including evidence limited to CT scan only.
* Brain metastases that have not been adequately treated with surgery or stereotactic radiosurgery and have not been stable at least 3 months prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To assess safety and tolerability during and for 1 hour following a 15 mg/kg dose of CP 675,206 administered as a one hour infusion. | Last patient dosed = 31Dec2009

SECONDARY OUTCOMES:
To monitor for human anti human (HAHA) response to CP 675,206 | Last HAHA time point obtain =estimated 31Dec2009
To assess evidence of anti tumor activity as measured by best overall response rate using Response Evaluation Criteria in Solid Tumors (RECIST) criteria, duration of response, progression free survival | Last RECIST obtained = estimated 31Dec2009
To identify potential relationships between polymorphisms in the Cytotoxic T lymphocyte associated antigen 4 (CTLA4), Fcgamma receptor IIa (FcgRIIa), IgG2a genes with safety and/or immune response of subjects treated with CP 675,206 | Last PG obtained = estimated 31Dec2009
To evaluate the overall safety and tolerability of CP 675,206 in this population | Last patient dosed = estimated 31Dec2009
To characterize the pharmacokinetics (PK) of CP 675,206 following a one hour infusion | Last PK timepoint obtained =estiamted 31Dec2009

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Research Site, Scottsdale, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Aurora, Colorado
  - Research Site, Atlanta, Georgia
  - Research Site, Indianapolis, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, Durham, North Carolina

REFERENCES:
- [Derived] Ribas A, Chesney JA, Gordon MS, Abernethy AP, Logan TF, Lawson DH, Chmielowksi B, Glaspy JA, Lewis K, Huang B, Wang E, Hsyu PH, Gomez-Navarro J, Gerhardt D, Marshall MA, Gonzalez R. Safety profile and pharmacokinetic analyses of the anti-CTLA4 antibody tremelimumab administered as a one hour infusion. J Transl Med. 2012 Nov 21;10:236. doi: 10.1186/1479-5876-10-236. PMID 23171508